CLINICAL TRIAL: NCT04840979
Title: Discovery and Validation of Genetic Variants Affecting Microglial Activation in Alzheimer's Disease With 11C-ER176
Brief Title: Discovery and Validation of Genetic Variants Affecting Microglial Activation in Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Philip De Jager, Weil-Granat Professor of Neurology, Columbia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAT2774; RF1AG070438 (NIH)
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: PET scan; Inflammation; Genetic testing; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Inflammation; Cognitive Dysfunction | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Impairment (Experimental): Subjects diagnosed with Alzheimer's disease (AD) or mild cognitive impairment (MCI) will have one PET scan with 11C-ER176, with arterial sampling. If the subject lacks known AD-biomarkers, they may undergo a 18F-florbetaben PET scan prior to the 11C-ER176 PET scan. Genome-wide genetic analysis will be performed. Participants will undergo an annual clinical evaluation and blood sample collection for 5 years to establish the trajectory of AD-related serum biomarkers and syndromic diagnoses.
  Interventions: Drug: 11C-ER176; Drug: 18F-florbetaben
- No Cognitive Impairment (Active Comparator): Healthy volunteers who are cognitively normal will have one PET scan with 11C-ER176, with arterial sampling. If the subject lacks known AD-biomarkers, they may undergo an 18F-florbetaben PET scan prior to the 11C-ER176 PET scan. Genome-wide genetic analysis will be performed. Participants will undergo an annual clinical evaluation and blood sample collection for 5 years to establish the trajectory of AD-related serum biomarkers and syndromic diagnoses.
  Interventions: Drug: 11C-ER176; Drug: 18F-florbetaben

INTERVENTIONS:
Drug: 11C-ER176 — 11C-ER176 is a novel TSPO radioligand that was developed because of its relative insensitivity to the rs6971 polymorphism. Increased TSPO signal on PET is associated with activation of microglia in the brain. The radioligand will be administered in tracer doses at activity of up to 20 mCi (740 MBq), IV, total of one injection. A single dose of radioligand will be injected over 1 minute.
  Other Names: [11C]ER176
Drug: 18F-florbetaben — Florbetaben has been approved by the FDA to help diagnose Alzheimer's disease. Florbetaben measures amyloid in the brain.
  Other Names: [18F] Florbetaben

SUMMARY:
The primary objectives are to validate that a previously identified gene variant influences the proportion of activated microglia (PAM) and the amount of TSPO binding on PET imaging, to identify novel loci that influence PAM and TSPO PET, and to understand the functional consequences of gene variants that drive microglial activation in Alzheimer's disease.

DETAILED DESCRIPTION:
While activated microglia have been observed in the vicinity of neuritic amyloid plaques in Alzheimer's disease (AD), there have been no large-scale assessments of microglial activation in aging and neurodegenerative disease. The investigators seek to understand the genetic underpinning of microglial responses-particularly the proportion of microglia in a morphologically-defined state of activation-that increase susceptibility to AD, so the investigators can develop more targeted forms of immune-based therapies to prevent cognitive decline and progression to dementia. The objective is to refine the genetic architecture of microglial activation to validate a previously identified gene variant -- and to identify novel loci -- that influence the proportion of activated microglia. The investigators also seek to understand the functional consequences of variants driving microglial activation in AD.

The central hypothesis is that identifiable gene variants influence microglial activation and susceptibility to AD. The investigators will test this hypothesis by conducting genome-wide analysis and identifying associations between gene variants and microglial activation. Microglial activation will be measured in human autopsy tissue (ex vivo), living human brain using PET imaging (in vivo), and in monocyte-derived microglia-like cells (in situ and in vitro).

This genetic study is designed to validate a finding that was discovered in participants with self-reported European-Caucasian ancestry. Therefore, the study seeks to enroll participants who self-report as white, not Hispanic or Latino. However, if this study is successful, the investigators plan to use the methods in this protocol in a future study to identify new genetic variants associated with changes on TSPO PET in a more diverse participant population. The investigators intend to use the results from this study to eventually benefit individuals of all racial and ethnic groups.

ELIGIBILITY:
Inclusion criteria:

1. Age 50 and older at time of study entry.
2. Meet criteria for either a) amnestic mild cognitive impairment (single or mixed domain) or Alzheimer's disease, or b) have no cognitive impairment, based on history, exam, and neuropsychological testing.
3. Patients must have Clinical Dementia Rating Scale score of 0.5 or 1 at enrollment. Controls must have Clinical Dementia Rating scale score of 0 at enrollment.
4. Subjects must have AD biomarker previously obtained for research or clinical purposes or undergo a 18F-florbetaben PET scan during the screening process. Patients must have positive amyloid PET scan or CSF results consistent with AD. Controls must have a negative amyloid PET scan or CSF results not consistent with AD.
5. Self-identify as white, non-Hispanic or Latino
6. Subjects must be ableto provide informed consent
7. Written and oral fluency in English
8. Able to participate in all scheduled evaluations and to complete all required tests and procedures.
9. In the opinion of the investigator, the subject must be considered likely to comply with the study protocol and to have a high probability of completing the study.

Exclusion Criteria:

1. Past or present history of certain brain disorders other than MCI or AD.
2. Certain significant medical conditions, which make study procedures of the current study unsafe. Such serious medical conditions include uncontrolled epilepsy and multiple serious injuries.
3. Contraindication to MRI scanning
4. Conditions precluding entry into the scanners (e.g. morbid obesity, claustrophobia, etc.).
5. Exposure to research related radiation in the past year that, when combined with this study, would place subjects above the allowable limits.
6. Participation in the last year in a clinical trial for a disease modifying drug for AD.
7. Inability to have a catheter in subject's vein for the injection of radioligand.
8. Inability to have blood drawn from subject's veins.
9. Taking anticoagulant (e.g., warfarin) or immunosuppressive/immunomodulatory medication. Nonsteroidal anti-inflammatory drugs (NSAIDs) are not exclusionary. Use of steroids in the 30 days preceding the PET scan.
10. Having a diagnosis of a chronic inflammatory disease (for example, multiple sclerosis, inflammatory bowel disease, rheumatoid arthritis, psoriasis, systemic lupus erythematosus) or a chronic infectious disease such as H.I.V.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between the chromosome 1 variant (rs2997325) and TSPO binding | Up to 1 year
  The measure will be in vivo validation of GWAS and assessment of clinical relevance by performing TSPO PET imaging using 11C-ER176 to measure microglial activation. PET images will be analyzed using 1) the two-tissue kinetic model to calculate total distribution volume, corrected for free fraction of radioligand in plasma (VT/fP). Analysis will be a meta-analysis of the association of rs2997325 with 11C-ER176 binding (total distribution volume, VT).
Number of variants discovered in genome-wide association study (GWAS) that influence TSPO binding | Up to 1 year
  11C-ER176 data will be used to perform a discovery GWAS for additional variants that influence TSPO binding and to define the genetic architecture of the PAM trait. Using PLINK and all imputed high quality genotypes (imputation r2 >0.8), adjusted for sex, age, and technical variables, the investigators will perform a GWAS for TSPO binding.

CONTACTS AND LOCATIONS:
Overall Officials: Philip De Jager, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available upon reasonable request from a qualified investigator.
Time Frame: Up to two weeks after review and approval of request.
Access Criteria: Investigator qualifications and previous work will be reviewed by PI. Subsequent email correspondence will relay technical criteria needed for access.